CLINICAL TRIAL: NCT02471794
Title: Personalized Health Planning in Shared Medical Appointments for Individuals With Type II
Brief Title: Personalized Health Planning in Shared Medical Appointments for Individuals With Type II Diabetes Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00063493
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Type II Diabetes
Keywords: Type II Diabetes; Personalized Health Planning; Shared Medical Appointments
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Shared Medical Appointment (No Intervention): The SMA group will be a standard shared diabetes medical appointment group consisting of up to 10 patients that utilizes the design and curriculum of the SMAs that are currently being held at the Duke Family Medicine Center.
- Personalized Health Planning Shared Medical Appointment (Experimental): The PHP SMA group will combine personalized health planning with a modified version of the standard shared diabetes medical appointment. Modifications include: a self-assessment of health status, greater emphasis on a collaborative patient-provider health goal-setting process, a plan to meet goals, a mindfulness practice included in each session, and the creation of a 'personalized health plan' participant notebook for each individual to document health goals and track progress to review at each session. The participant notebook also includes educational handouts and worksheets to complement the educational curriculum.
  Interventions: Behavioral: Personalized Health Planning Shared Medical Appointment
- Retrospective (No Intervention): A retrospective chart review will be conducted once all participants (both SMA group and PHP SMA group) complete the intervention. The retrospective chart review will collect healthcare utilization data six months prior, during, and after each subject's participation in the SMA.

INTERVENTIONS:
Behavioral: Personalized Health Planning Shared Medical Appointment — The PHP SMA group will combine personalized health planning with a modified version of the standard shared diabetes medical appointment. Modifications include: a self-assessment of health status, greater emphasis on a collaborative patient-provider health goal-setting process, a plan to meet goals, a mindfulness practice included in each session, and the creation of a 'personalized health plan' participant notebook for each individual to document health goals and track progress to review at each session. The participant notebook also includes educational handouts and worksheets to complement the educational curriculum
  Arms: Personalized Health Planning Shared Medical Appointment

SUMMARY:
The primary aim of this study is to examine the feasibility of implementing an evidence based patient engagement strategy, known as personalized health planning (PHP), in the context of a a shared medical appointment (SMA) for individuals with type II diabetes in a primary care setting.

DETAILED DESCRIPTION:
All data for the prospective portion of this study was done being collected in September 2016. The retrospective chart review will collect data up until March of 2017 (six months after the last subject completed the prospective phase by attending their last SMA session).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Type 2 diabetes within the last year
* A current patient at Duke Family Medicine.
* An A1C score greater than 7 and less than 14.

Exclusion Criteria:

* A diagnosis of Pre-diabetes
* A diagnosis of Type I diabetes
* Individuals with amputations as a result of their diabetes are excluded form this study.
* Individuals with renal dialysis will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Feasibility measured using a patient satisfaction survey | 12 months
Change in patient activation measured using the patient activation measure | baseline; 6 months; 12 months
Change in self-management of diabetes self-efficacy using the Diabetes Empowerment Scale | baseline; 6 months; 12 months
Change in diabetes self efficacy using the 1-item diabetes self-efficacy scale | baseline; 6 months; 12 months
Change in A1C using the A1C blood test | baseline; 3 months; 6 months; 9 months; 12 months

SECONDARY OUTCOMES:
Change in depression screening score using the Patient Health Questionnaire (PHQ-9) | baseline; 6 months; 12 months
Change in functional health and well-being using the short form health survey | baseline; 6 months; 12 months
Change in general self-rated health using the general self rated health survey (GSRH) | baseline; 6 months; 12 months
Change in health goal progress using a goal progress visual analog scale | 3 months; 10 months
change in body mass index using weight and height measurements | baseline; 1 months; 2 months; 3 months; 5 months; 8 months; 10 months; 12 months
change in blood pressure using blood pressure measurement | baseline; 1 months; 2 months; 3 months; 5 months; 8 months; 10 months; 12 months
Change in low-density lipoprotein cholesterol (LDL) using LDL measurement | baseline; 6 months; 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hull, MD MPH, Principal Investigator — Duke University
Locations (1):
- Duke Family Medicine Center, Durham, North Carolina, United States